CLINICAL TRIAL: NCT06246565
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-designed Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of HS-10383 in Chinese Adult Subjects With Refractory or Unexplained Chronic Cough (RUCC)
Brief Title: A Study of HS-10383 in Chinese Adult Subjects With Refractory or Unexplained Chronic Cough (RUCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10383-201
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-01

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-10383 50mg (Experimental): HS-10383 oral dose 50 mg once a day.
  Interventions: Drug: HS-10383
- HS-10383 100mg (Experimental): HS-10383 oral dose 100 mg once a day.
  Interventions: Drug: HS-10383
- HS-10383 200ng (Experimental): HS-10383 oral dose 200 mg once a day.
  Interventions: Drug: HS-10383
- Placebo (Placebo Comparator): Matching Placebo for HS-10383 oral dose once a day
  Interventions: Drug: HS-10383 Placebo

INTERVENTIONS:
Drug: HS-10383 — HS-10383 administered as one 50 mg, 100 mg 200 mg tablet once daily, depending upon randomization.
  Arms: HS-10383 100mg; HS-10383 200ng; HS-10383 50mg
Drug: HS-10383 Placebo — HS-10383 administered as one 50 mg, 100 mg 200 mg tablet once daily, depending upon randomization.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-designed phase 2 clinical trial to evaluate the efficacy, safety and pharmacokinetic (PK) characteristics of HS-10383 in Chinese adult subjects with refractory or unexplained chronic cough (RUCC).

DETAILED DESCRIPTION:
The primary objectives of this study are to evaluate the efficacy of HS-10383 in reducing cough frequency as measured over a 24-hour period, and to determine the safety and tolerability of HS-10383. The primary hypothesis is that at least one dose of HS-10383 is superior to placebo in reducing coughs per hour (over 24 hours) at Week 4.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should have a full understanding of the study contents, process, and possible adverse reactions, and voluntarily sign the informed consent form;
2. Subjects aged 18-70 years (including the critical value) with RUCC ≥1 year (diagnosis of RUCC according to the Expert Consensus on Diagnosis and Treatment of Refractory Chronic Cough in China [Released in 2021]);
3. Subjects whose serum pregnancy test is negative in both screening and baseline visits;

Exclusion Criteria:

1. Subjects who are diagnosed with chronic obstructive pulmonary disease, bronchiectasis, idiopathic pulmonary fibrosis and other serious lung diseases;
2. Any physiological or mental disease or condition that may increase study risks or interfere with the conduct of the study or affect the ability to complete this study in the opinion of the investigator, such as medical history of depression;
3. Subjects who cannot meet the requirements for piror treatment or who cannot adhere to the concomitant treatment as specified in Section 6.7-Prior/concomitant medications and non-drug treatment.
4. Subjects with positive hepatitis A IgM antibody, hepatitis C antibody (HCVAb), syphilis antibody or human immunodeficiency virus (HIV) antibody at screening visit; subjects with positive hepatitis B surface antigen (HBsAg) at screening (except for quantitative detection result of HBV-DNA is below the lower limit of the detection reference range).
5. Any former smoker with more than 20 packs/year; or have quited smoking for less than 6 months; or subjects who are still smoking (including e-cigarettes);
6. Subjects who have a history of serious drug, food or environmental allergies, or who are known to be allergic to the ingredients of investigational product;
7. History of drug dependence,drug or alcohol abuse in the past year;
8. Female subjects who are pregnant or breastfeeding;
9. Subjects who have previously received anything that may affect drug absorption, including but not limited to: gastrectomy, gastroplasty, any type of weight-loss surgery, vagotomy or enterotomy;
10. Subjects who have been vaccinated within 30 days before screening visit, or have a vaccination plan during the whole study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
24-Hour Cough Frequency | at Week 4
  Assessed using an ambulatory cough monitor

SECONDARY OUTCOMES:
Awake Cough Frequency | at Week 4
  Change from baseline in awake cough frequency at week 4;
Change from Baseline in Cough Severity Visual Analogue Scale at Week 2 and Week 4; | at Week 2 and Week 4
  Assessed by Cough Severity Visual Analogue Scale [VAS] by the participant on a 100 mm visual analog scale where higher scores indicate greater severity.
Change from Baseline in the Leicester Cough Questionnaire (LCQ) Total Score at Week 2 and Week 4. | at Week 2 and Week 4
  The LCQ is a patient-reported quality of life (QOL) measure of chronic cough，the higher scores mean a better outcome.